CLINICAL TRIAL: NCT04912583
Title: Comparison of Mechanical Ventilation With Low and High Tidal Volumes in Acute Spinal Cord Injury: A Pilot Randomized Comparative Effectiveness Trial
Brief Title: Comparison of Low and High Tidal Volumes in Acute Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: TIRR Memorial Hermann (Other); Craig Hospital (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Radha Korupolu, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-21-0222; KL2TR003168 (NIH)
Record Dates: First submitted 2021-04-29; First posted 2021-06-03 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury; Mechanical ventilation; Pneumonia; Tidal volume
MeSH Terms: conditions — Spinal Cord Injuries; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, principal investigator, outcome assessors, and statistician will be blinded to tidal volume assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High tidal volume (Active Comparator): A high tidal volume (14-16 ml/kg pbw) with positive end-expiratory pressure will be applied during mechanical ventilation.
  Interventions: Device: High tidal volume
- Low tidal volume (Active Comparator): A low tidal volume (8-10 ml/kg pbw) with positive end-expiratory pressure will be applied during mechanical ventilation.
  Interventions: Device: Low tidal volume

INTERVENTIONS:
Device: High tidal volume — A high tidal volume (14-16 ml/kg pbw) with positive end-expiratory pressure will be applied during mechanical ventilation.
  Arms: High tidal volume
Device: Low tidal volume — A low tidal volume (8-10 ml/kg pbw) with positive end-expiratory pressure will be applied during mechanical ventilation.
  Arms: Low tidal volume

SUMMARY:
Objective: This study's primary objective is to evaluate the efficacy and feasibility of mechanical ventilation with high vs. low tidal volume (Vt) in people with acute spinal cord injury (SCI). Secondary objectives include a comparison of inflammatory markers between these groups.

Study Design: Randomized comparative effectiveness trial

Methods: Study population: Adults with acute traumatic SCI on mechanical ventilation (MV). Subjects will be randomized to receive either a lower Vt of 8-10 cc/kg predicted body weight (pbw) or a high Vt of 14-16 ml/kg pbw.

Risks and potential Benefits: Risks of study interventions are similar to usual care as proposed tidal volume settings are within the current usual care range. However, people assigned to the lower tidal volume group may have a lower risk of pneumonia and respiratory complications.

DETAILED DESCRIPTION:
Background: Respiratory complications associated with mechanical ventilation (MV) are the leading cause of morbidity and mortality following acute spinal cord injury (SCI). Emerging evidence suggests pneumonia is also associated with reduced neurologic recovery. Therefore, pneumonia prevention is of primary importance to improve outcomes. In the non-SCI population, MV with lower tidal volume (Vt) has been shown to reduce inflammation and rates of pneumonia. High Vt MV results in disruption of pulmonary endothelium and release of inflammatory mediators, which play a role in the development of pulmonary complications. In contrast, guidelines for SCI practitioners recommend MV with higher Vt without strong evidence.

Objective: The primary objective of this study is to evaluate the feasibility of conducting a randomized control trial comparing MV with high vs. low Vt. Secondary objectives include a comparison of clinical outcomes and inflammatory mediators between these groups.

Methods: Study population: Adults with acute traumatic SCI admitted to an acute inpatient rehabilitation facility on MV. Subjects will be randomized to receive either a lower Vt of 8-10 cc/kg predicted body weight (pbw) or a high Vt of 14-16 ml/kg pbw. Study participants will be randomly assigned to high tidal volume (14-16 ml/kg pbw) or low tidal volume of 8 to 10 ml/kg pbw within 48 hrs of admission, stratified based on vital capacity at admission to ensure equal allocation of those with most severe respiratory impairment and unlikely to wean from the vent.

Importance of knowledge gained from the study: Investigators believe the completion of this study will add to the fund of knowledge of respiratory management of people with SCI, especially at the early stages of the injury, including reducing respiratory complications in people with SCI who are at very high risk of severe respiratory complications which is the main cause of morbidity and mortality in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years (Lung volumes and ventilator settings are different for ages <18 years).
* Acute SCI of duration ≤ four months
* Mechanical ventilation subjects: traumatic or non-traumatic cervical SCI with neurological level C1-C5 admitted to our acute inpatient rehabilitation facility (AIR) on mechanical ventilation

Exclusion Criteria:

* Severe dysphagia due to concomitant brain stem injury, which increases the risk of pneumonia
* Severe brain injury resulting in dysphagia and inability to follow instructions to perform vital capacity measurements
* ARDS or severe lung disease (required supplemental oxygen or ventilator prior to SCI) at the time of admission (these conditions will not allow patients to randomize because target vt may below)
* Prolonged antibiotics for > 3 weeks at the time of admission due to infection (e.g., osteomyelitis, epidural abscess, etc.),
* Presence of diaphragmatic pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radha Korupolu, MD, Principal Investigator — McGovern Medical School, The University of Texas Health Science Center at Houston
Locations (2):
- United States (2):
  - Craig Hospital, Englewood, Colorado
  - TIRR Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hatton GE, Mollett PJ, Du RE, Wei S, Korupolu R, Wade CE, Adams SD, Kao LS. High tidal volume ventilation is associated with ventilator-associated pneumonia in acute cervical spinal cord injury. J Spinal Cord Med. 2021 Sep;44(5):775-781. doi: 10.1080/10790268.2020.1722936. Epub 2020 Feb 11. PMID 32043943
- [Background] Korupolu R, Stampas A, Uhlig-Reche H, Ciammaichella E, Mollett PJ, Achilike EC, Pedroza C. Comparing outcomes of mechanical ventilation with high vs. moderate tidal volumes in tracheostomized patients with spinal cord injury in acute inpatient rehabilitation setting: a retrospective cohort study. Spinal Cord. 2021 Jun;59(6):618-625. doi: 10.1038/s41393-020-0517-4. Epub 2020 Jul 9. PMID 32647326

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 62 participants were screened for eligibility. Of those, 31 met the inclusion criteria and signed informed consent. One participant was transferred before randomization and did not continue in the study. A total of 31 participants were enrolled, and 30 were randomized.
Period: Overall Study
Arm/Group | High Tidal Volume | Low Tidal Volume
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Tidal Volume | High Tidal Volume | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Standard Deviation); unit: years] | 54 (13) | 44 (17) | 49 (15.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Cause of injury [Count of Participants; unit: Participants]
  Vehicular | 8 | 7 | 15
  Fall | 4 | 3 | 7
  Violence | 1 | 1 | 2
  Medical/Surgical Complications | 1 | 0 | 1
  Sports | 1 | 3 | 4
  Other traumatic Injuries | 0 | 1 | 1
Asia Impairment Scale Classification [Count of Participants; unit: Participants] — The Asia Impairment Scale (AIS) categorizes spinal cord injury severity based on sensory and motor function loss.
  AIS Classification:
  A = Complete: No motor/sensory function in the sacral segments S4-S5 B = Incomplete: Sensory but not motor function below the neurological level, includes the sacral segments S4-S5 C = Incomplete: Below the neurological level, motor function preserved and more than 50% of key muscles have a muscle grade < 3 D = Incomplete: Below the neurological level, motor function persevered and at least 50% of key muscles have a muscle grade ≥3
  Participants
    A | 9 | 11 | 20
    B | 5 | 2 | 7
    C | 1 | 2 | 3
    D | 0 | 0 | 0
Number of Participants with a smoking history [Count of Participants; unit: Participants] | 5 | 3 | 8
Number of participants with a history of lung or pulmonary disorders prior to Spinal Cord Injury [Count of Participants; unit: Participants] | 0 | 1 | 1
Number of participants with a history of concomitant mild traumatic brain injury or stroke [Count of Participants; unit: Participants] | 5 | 2 | 7
Neurological Level of Spinal Cord Injury (SCI) [Count of Participants; unit: Participants] — Neurological Level of Spinal Cord Injury was measured by the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) exam. ISNCSCI exam provides an overall assessment of motor and sensory function following spinal cord injury. Participants were grouped into the following categories:
  C1-C3: High cervical injuries; individuals typically require ventilator support for a prolonged duration.
  C4-C5: Mid-cervical injuries, who may require ventilator support for a shorter duration following SCI.
  Participants
    C1 to C3 | 7 | 9 | 16
    C4 to C5 | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Episodes of Pneumonia
Description: The primary outcome is pneumonia episodes with evidence of new or progressive and persistent infiltrate on chest radiograph plus 2 of the following abnormal white blood cell count, presence of fever or hyperthermia, purulent sputum, and deterioration in gas exchange. Any new pneumonia episodes which meet the above criteria and developed 48 hours after achieving target tidal volume will be recorded.
Time Frame: From the time of enrollment to time of discharge from hospital (about 6 weeks)
Measure: Mean (Standard Deviation); unit: episodes of pneumonia
Arm/Group | High Tidal Volume | Low Tidal Volume
Number analyzed (Participants) | 15 | 15
episodes of pneumonia | .13 (.35) | .4 (.5)

2. Secondary Outcome: Feasibility as Assessed by Recruitment Rate
Description: Recruitment rate is the proportion of eligible people who provide consent.
Time Frame: At the time of consent (within 48 hours of hospital admission)
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Screened: All subjects who were screened
Arm/Group | All Subjects Screened
Number analyzed (Participants) | 62
Participants | 31

3. Secondary Outcome: Feasibility as Assessed by Adherence Rate
Description: Adherence rate is the proportion of participants in each group who receive the assigned intervention per protocol.
Time Frame: At the time of start of intervention (within 48 hours of hospital admission)
Measure: Count of Participants; unit: Participants
Arm/Group | High Tidal Volume | Low Tidal Volume
Number analyzed (Participants) | 15 | 15
Participants | 11 | 13

4. Secondary Outcome: Feasibility as Assessed by Retention Rate
Description: Retention rate is the number of participants in each group who complete all study procedures.
Time Frame: at the time of discharge from hospital (about 6 weeks after admission)
Measure: Count of Participants; unit: Participants
Arm/Group | High Tidal Volume | Low Tidal Volume
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

5. Secondary Outcome: Feasibility as Assessed by Number of Participants With Missing Data
Time Frame: From the time of enrollment to time of discharge from hospital (about 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Low Tidal Volume | High Tidal Volume
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

6. Other Pre Specified Outcome: Number of Respiratory Complications
Description: The following ventilator-associated events will be reported: transfer to acute care hospital due to respiratory complications, weaning failure, new pneumothorax, Acute respiratory distress syndrome (ARDS), pleural effusion, pulmonary embolism, atelectasis, and pulmonary edema.
Time Frame: From the time of enrollment to the time of discharge from the hospital (about 6 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of enrollment to time of discharge from hospital (about 6 weeks)
Arm/Group | High Tidal Volume | Low Tidal Volume
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 12/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Tidal Volume (N=15) | Low Tidal Volume (N=15)
Cardiac Arrest (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Tidal Volume (N=15) | Low Tidal Volume (N=15)
Urinary tract infection (Renal and urinary disorders) | 8 | 6
Sacral Wound Infection (Infections and infestations) | 2 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Vaginal Infection (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Mucus plug, which required a transfer (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis/Tracheitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Atelectasis requiring intervention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COVID (General disorders) | 1 | 1
Pneumonia after 48 hours of admission (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT04912583/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT04912583/ICF_001.pdf